CLINICAL TRIAL: NCT06822062
Title: The Effect of Chitin and Ascorbic Acid on Dietary Iron Absorption From Tenebrio Molitor Larvae in Young Women.
Brief Title: Effect of Chitin and Ascorbic Acid on Dietary Insect Iron Absorption
Acronym: INSECTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Distance University of Applied Sciences (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: INSECTE_01
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiency (Without Anemia)
Keywords: edible insects; Tenebrio molitor; iron deficiency; iron bioavailability; chitin; ascorbic acid
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: The study will be a single-center, prospective cross-over trial, in which all study participant will receive the seven test conditions.
Who Masked: Participant
Masking Description: The randomization will be single-blinded, i.e., the participants will not know which type of test meal they will be given on which study visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- T.molitor native chitin (Experimental): Vegetable soup prepared with dried 57-Fe intrinsically labeled T.molitor
  Interventions: Other: Meal A
- T.molitor high chitin level (Experimental): Vegetable soup prepared with dried 57-Fe intrinsically labeled T.molitor + 2g chitin of shrimp origin
  Interventions: Other: Meal B
- T.molitor + Ascorbic Acid (Experimental): Vegetable soup prepared with dried 57-Fe intrinsically labeled T.molitor + Ascorbic acid (4:1 ascorbic acid to iron molar ratio)
  Interventions: Other: Meal C
- Control meal (Experimental): Vegetable soup with addition of labelled FeSO4 (isotope iron 58)
  Interventions: Other: Meal D
- Control meal low chitin (Experimental): Vegetable soup with addition of labelled FeSO4 (isotope iron 58) + 1g chitin of shrimp origin
  Interventions: Other: Meal E
- Control meal high chitin (Experimental): Vegetable soup with addition of labelled FeSO4 (isotope iron 58) + 3g chitin of shrimp origin
  Interventions: Other: Meal F
- Control meal + Ascorbic Acid (Experimental): Vegetable soup with addition of labelled FeSO4 (isotope iron 54) + Ascorbic acid (4:1 ascorbic acid to iron molar ratio)
  Interventions: Other: Meal G

INTERVENTIONS:
Other: Meal A — Vegetable soup prepared with dried intrinsically labeled T.molitor (isotopic iron 57, native chitin content = 1g)
  Arms: T.molitor native chitin
Other: Meal B — Vegetable soup prepared with dried intrinsically labeled T.molitor (isotopic iron 57) + 2g of extrinsically added chitin
  Arms: T.molitor high chitin level
Other: Meal C — Vegetable soup prepared with dried intrinsically labeled T.molitor (isotopic iron 57) + ascorbic acid (4:1 ascorbic acid to iron molar ratio)
  Arms: T.molitor + Ascorbic Acid
Other: Meal D — Vegetable soup without insects with extrinsic addition of FeSO4 (isotopic iron 58)
  Arms: Control meal
Other: Meal E — Vegetable soup without insects with extrinsic addition of FeSO4 (isotopic iron 58) + 1g of extrinsically added chitin
  Arms: Control meal low chitin
Other: Meal F — Vegetable soup without insects with extrinsic addition of FeSO4 (isotopic iron 58) + 3g of extrinsically added chitin
  Arms: Control meal high chitin
Other: Meal G — Vegetable soup without insects with extrinsic addition of FeSO4 (isotopic iron 54) + ascorbic acid (4:1 ascorbic acid to iron molar ratio)
  Arms: Control meal + Ascorbic Acid

SUMMARY:
Iron is involved in many vital metabolic processes such as oxygen transport, electron transport in cells, DNA synthesis and repair, and muscle metabolism. However, iron deficiency and iron deficiency anemia continue to affect many people, particularly preschool children (<5 years), adolescents, and pregnant and non-pregnant women of childbearing age. Iron deficiency is characterized by a lack of total iron stores in the body, which is mainly caused by insufficient dietary iron intake, physiologically increased iron requirements, poor intestinal iron absorption, or chronic blood loss. Animal foods are important sources of highly bioavailable iron in the human diet. Meeting human nutritional needs for the rapidly increasing world population while targeting food production within the planetary boundaries will require the identification of sustainable iron sources, such as edible insects. A previous iron absorption study showed that insect iron is absorbed moderately well. The present study will examine if and to which extent chitin, a polysaccharide within the insect biomass, inhibits iron absorption. In addition, the enhancing iron absorption of ascorbic acid on iron absorption from Tenebrio molitor larvae will be studied. This knowledge can support to optimize the composition of an insect-based meal to increase its iron absorption.

To distinguish iron absorption from insect biomass from other sources, insects are labeled with stable iron isotopes (Fe-57, Fe-58, Fe-54) and iron absorption in the blood is measured.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 18-45 years
* Normal BMI (18.5 - 24.9 kg/m2)
* Body weight < 70 kg
* Low iron status (being in the lower half of the serum ferritin distribution at screening)

Exclusion Criteria:

* Anaemia (Hb < 12 g/dL)
* Inflammation (CRP > 5.0 mg/L)
* Pregnancy or intention to become pregnant during the study or within 30 days after the discontinuation of the study intervention
* Lactating up to 6 weeks before the study initiation
* Chronic digestive, renal and/or metabolic diseases
* Antibiotics in the last 4 weeks prior to the study and during the study
* Mineral and vitamin supplementation in the last 2 weeks prior to the study and during the course of the study
* Chronic medication intake (except for oral contraceptives)
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Earlier participation in a study using stable isotopes or in any clinical study within the last 30 days
* Food allergies, especially known hypersensitivity to crustacea, dust mites, sea food, gluten, milk, or eggs
* Cigarette smoking (> 1 cigarette per day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fractional iron absorption | screening (-1), 16th, 32nd,47th day of the study
  Fractional iron absorption will be calculated based on the shift in iron isotope ratio in red blood cells 14 to 16 days post administration of the isotopically labelled meals. Calculation of fractional iron absorption will take into account the principles of isotope dilution and the fact that iron isotopic labels are not monoisotopic.

SECONDARY OUTCOMES:
Hemoglobin (Hb) | screening (-1), 16th, 32nd, 47th day of the study
  Iron status marker
Serum Ferritin (SF) | screening (-1), 16th, 32nd, 47th day of the study
  Iron status marker
Serum Transferrin Receptor (sTfR) | screening (-1), 47th day of the study
  Iron status marker
C-Reactive Protein (CRP) | screening (-1), 16th, 32nd, 47th day of the study
  Inflammation status
alpha-1-acid glycoprotein (AGP) | screening (-1), 47th day of the study
  Inflammation status
Retinol binding Protein (RBP) | screening (-1), 47th day of the study
  Inflammation status

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, Prof., Principal Investigator — Fernfachhochschule Schweiz
Locations (1):
- ETH Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided